CLINICAL TRIAL: NCT06033001
Title: Expanded Access Treatment with [Lu-177]-PNT2002 for Adult Patients with Prostate-Specific Membrane Antigen (PSMA)-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Temporarily not available | Type: Expanded Access
Sponsor: Lantheus Medical Imaging (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: LNTH-PNT2002-EAP01
Record Dates: First submitted 2023-08-10; First posted 2023-09-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Castration-Resistant Prostatic Cancer
Keywords: progressive mCRPC
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: [Lu-177]-PNT2002 — [Lu-177]-PNT2002, is a radiopharmaceutical investigational drug. [Lu-177]-PNT2002 targets a specific protein that is located on the surface of prostate cancer cells called PSMA. [Lu-177]-PNT2002 delivers radiation to your cancer by binding to the PSMA which helps destroy the cancer cells. [Lu-177]-PNT2002 is administered intravenously every 8 weeks (about every 2 months) for 4 cycles, or 8 months of total treatment.

SUMMARY:
The purpose of this program is to provide access to [Lu-177]-PNT2002 to patients who have been diagnosed with prostate-specific membrane antigen (PMSA)-positive castration-resistant prostate cancer (mCRPC). Patients must have received at least 1 prior androgen pathway inhibitor (ARPI) and cannot be treated by currently available drugs or clinical trials.

In this program participants will be administered [Lu-177]-PNT2002 intravenously every 8 weeks (about every 2 months) for 4 cycles, or 8 months of total treatment. During treatment, participants will be monitored with routine laboratory tests such as:

* Hematology blood tests
* Clinical Chemistry blood tests
* Testosterone/Prostate Antigen levels blood test
* Vital signs
* Imaging
* ECG

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male aged 18 years or older;
2. Histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate;
3. Patients must have at least 1 metastatic lesion present on CT, MRI, or bone scan imaging;
4. Patients must have progressive mCRPC based on at least 1 of the following criteria:

   1. Serum/plasma PSA progression defined as increase in PSA greater than 25% and >2 ng/mL above nadir, confirmed by progression at 2 time points at least 3 weeks apart
   2. Soft-tissue progression defined as an increase ≥20% in the sum of the diameters (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or a new lesion
   3. Progression of bone disease defined as the appearance of 2 or more lesions by bone scan
5. Progression on prior treatment with ≥1 ARPI (abiraterone, apalutamide, darolutamide, enzalutamide ) in nmCRPC, mHSPC or mCRPC;
6. PSMA-PET scan ([Ga-68]-PSMA-11 or [F-18]-DCFPyL) positive as determined by local investigator;

   1. At least 1 PSMA-PET positive lesion for prostate cancer
   2. Uptake greater than the liver will be used as the reference for determining PSMA-PET positivity and uptake less than or equal to the liver will be used as the reference for determining PSMA-PET negativity
   3. All lymph nodes that measure ≥25 mm in short axis on anatomic imaging must be PSMA-PET positive
   4. All bone metastases with soft tissue component(s) ≥10 mm in short axis must be PSMA-PET positive (PSMA-negative osseous metastases without a soft tissue component do not exclude patients)
   5. All solid organ metastases (i.e., lung, liver, adrenal glands, etc.) ≥10 mm in short axis must be PSMA-PET positive
7. Castrate levels of circulating testosterone (<1.7 nmol/L or <50 ng/dL);
8. Patients must have recovered to Grade ≤2 from all clinically significant toxicities related to; prior therapies (i.e., prior ARPI, chemotherapy, PARPi, radioisotope or immunotherapy, etc.)
9. Adequate organ function, independent of transfusion;

   a. Bone marrow reserve

   i. White blood cell (WBC) count ≥2.5 x 109/L OR absolute neutrophil count (ANC) ≥1.5 x 109/L ii. Platelets ≥100 x 109/L iii. Hemoglobin ≥80 g/L or ≥8 g/dL

   b. Liver function

   i. Total bilirubin ≤1.5 x institutional upper limit of normal (ULN). For patients with known Gilbert's syndrome, ≤3.0 x ULN ii. ALT and AST ≤3.0 x ULN

   c. Renal function

   i. Creatinine clearance ≥50 mL/min based on Cockroft-Gault formula

   d. Albumin ≥30 g/L
10. Human immunodeficiency virus-infected patients who are healthy and have a low risk of acquired immunodeficiency syndrome-related outcomes are eligible;
11. ECOG performance status 0 or 1;
12. For patients who have partners who are pregnant or of childbearing potential: a condom is required along with a highly effective contraceptive method during the study and for 6 months after last study drug administration. Such methods deemed highly effective include a) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, b) progestogen-only hormonal contraception associated with inhibition of ovulation, c) intrauterine device (IUD), d) intrauterine hormone-releasing system (IUS), e) bilateral tubal occlusion, f) vasectomy, g) true sexual abstinence: when this is in line with the preferred and usual lifestyle of the subject [periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of abstinence].
13. Signed Informed Consent Form

Exclusion Criteria:

1. Prior PSMA-targeted radioligand therapy (i.e., [Lu-177]-PSMA-617);
2. A superscan defined as a bone scan that demonstrates markedly increased skeletal radioisotope uptake relative to soft tissues in association with absent or faint genitourinary tract activity;
3. Patients with a history of central nervous system (CNS) metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity;
4. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history or CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast);
5. Symptomatic cord compression, or clinical radiologic findings indicative of impending cord compression;
6. Any pre-existing symptoms, or concurrent severe and/or uncontrolled medical conditions such as ureteral obstruction, which in the opinion of the investigator would compromise safe participation in the [Lu-177]-PNT2002 EAP;
7. Not able to understand and comply with treatment instructions and requirements;

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Hartford HealthCare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - Florida Theranostics Cancer Center, Jupiter, Florida
  - Biogenix Molecular, LLC, Miami, Florida
  - Comprehensive Hematology Oncology, Trinity, Florida
  - BAMF Health, Inc, Grand Rapids, Michigan
  - John Theurer Cancer Center at Hackensack Meridian University Medical Center, Hackensack, New Jersey